CLINICAL TRIAL: NCT00899548
Title: DNA Methylation in Serum as a Predictive Marker of Progression and Survival Following Systemic Therapy in Patients With Metastatic Breast Cancer
Brief Title: DNA in Predicting Response After Systemic Therapy in Women With Metastatic Breast Cancer
Status: Completed | Type: Observational
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: J0524; P30CA006973 (NIH); JHOC-J0524 (Other: SKCCC at Johns Hopkins); JHOC-SKCCC-J0524 (Other: SKCCC at Johns Hopkins); CDR0000509417 (Other: NCI PDQ); NA_00000717 (Other: JHM IRB)
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Results first posted 2019-07-26 (Actual); Last update posted 2019-07-26 (Actual); Status verified 2019-07

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — DNA Methylation; Microarray Analysis; Polymerase Chain Reaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, plasma, DNA, RNA, whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Metastatic breast cancer patients: DNA methylation analysis, microarray analysis, polymerase chain reaction, laboratory biomarker analysis
  Interventions: Genetic: DNA methylation analysis; Genetic: microarray analysis; Genetic: polymerase chain reaction; Other: laboratory biomarker analysis

INTERVENTIONS:
Genetic: DNA methylation analysis — laboratory analysis
Genetic: microarray analysis — laboratory analysis
Genetic: polymerase chain reaction — laboratory analysis
Other: laboratory biomarker analysis — laboratory analysis

SUMMARY:
RATIONALE: Studying samples of blood from patients with cancer and from healthy participants in the laboratory may help doctors learn more about changes that may occur in DNA and identify biomarkers related to cancer. It may also help doctors predict how well patients will respond to systemic therapy.

PURPOSE: This laboratory study is looking at DNA in predicting response after systemic therapy in women with metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Identify a panel of methylated gene markers in serum from women with metastatic breast cancer that is significantly different from that observed in healthy participants.
* Assess changes in a panel of methylated gene markers from baseline, after 3-4 weeks, and after 9-12 weeks of systemic therapy in patients with metastatic breast cancer.
* Determine the potential effects of common exposures (i.e., alcohol, smoking, medications, and dietary factors) on patterns of serum methylation in patients with metastatic breast cancer and in healthy participants.
* Develop a predictive model using DNA methylation profiles in serum that predicts clinical outcome for an individual patient with metastatic disease.

Secondary

* Correlate circulating tumor cells (CTCs) with clinical outcome in patients with metastatic breast cancer.
* Correlate CTCs with serum methylation in these patients.
* Determine if the addition of CTCs to serum methylation results in an improved predictive model.

OUTLINE: This is a prospective, multicenter study.

Patients and healthy participants fill out health assessment questionnaires at baseline, week 3-4, and week 9-12.

Patients undergo blood collection for methylated marker analysis at baseline, weeks 3-4, and weeks 9-12 and circulating tumor cell levels at baseline and weeks 3-4. Healthy participants undergo blood collection for methylated marker analysis at baseline. An additional cohort of healthy participants undergo follow-up blood collection ≥ 1 week after baseline.

DNA methylation is measured by quantitative multiplex methylation-specific polymerase chain reaction (QM-MSP) assay.

After completion of study procedures, patients are followed every 3-4 months.

PROJECTED ACCRUAL: A total of 150 patients and 150 healthy participants will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Meets 1 of the following criteria:

  * Histologically and/or cytologically confirmed stage IV adenocarcinoma of the breast (patient)
  * No diagnosis of an abnormal breast biopsy (including atypical ductal or lobular hyperplasia), or new diagnosis of breast cancer or breast cancer recurrence within the past five years (healthy participant)
* Evidence of disease progression AND initiating a new systemic treatment regimen with trastuzumab (Herceptin®), chemotherapy, endocrine therapy, or investigational agent(s) (patient)

  * Treatment may be given as a single agent or in combination
* Measurable or evaluable disease (patient)

  * Measurable disease is defined as ≥ 1 measurable lesion identified by RECIST criteria
  * Patients with evaluable disease only must have ≥ 1 tumor marker (e.g., carcinoembryonic antigen, CA 27-29, or CA 15-3) above normal level
* Treated brain metastases (surgery or radiation therapy) allowed provided patient has evidence of disease stability or presence of other site(s) of measurable or evaluable disease (patient)

  * No leptomeningeal disease
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Female
* Menopausal status not specified
* ECOG performance status 0-2
* No known cancer within the past 5 years other than basal cell or squamous cell carcinoma of the skin and/or adequately treated cervical cancer (healthy participant)
* Not pregnant or nursing

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Prior therapy in the preoperative, adjuvant, and/or metastatic setting allowed

  * Any number of prior regimens in any setting allowed
* No prior radiation therapy to the only site of disease unless there is evidence of post-radiation disease progression
* No selective estrogen receptor modulator or aromatase inhibitor for breast cancer prevention or therapy within the past 12 months (healthy participant)
* Prior or concurrent use of raloxifene for osteopenia or osteoporosis therapy allowed (healthy participant)
* Concurrent participation in another clinical trial, including one involving an investigational agent(s), allowed

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Metastatic breast cancer patients and women without a history of breast cancer (ie, healthy women or "normals')
Sampling Method: Probability Sample
Enrollment: 182 (Actual)
Dates: Start 2007-01 (Actual); Primary Completion 2010-06 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antonio C. Wolff, MD, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (4):
- United States (4):
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina

IPD SHARING:
Plan to Share IPD: Yes
Data set will be available upon review and approval by the Correlative Science Review Committee of the Translational Breast Cancer Research Consortium (TBCRC). Inquiries should be addressed to the study chair, Dr. Antonio Wolff
Time Frame: Not yet determined
Access Criteria: Not yet determined

REFERENCES:
- [Result] Visvanathan K, Fackler MS, Zhang Z, Lopez-Bujanda ZA, Jeter SC, Sokoll LJ, Garrett-Mayer E, Cope LM, Umbricht CB, Euhus DM, Forero A, Storniolo AM, Nanda R, Lin NU, Carey LA, Ingle JN, Sukumar S, Wolff AC. Monitoring of Serum DNA Methylation as an Early Independent Marker of Response and Survival in Metastatic Breast Cancer: TBCRC 005 Prospective Biomarker Study. J Clin Oncol. 2017 Mar;35(7):751-758. doi: 10.1200/JCO.2015.66.2080. Epub 2016 Nov 21. PMID 27870562

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at each of the participating institutions at Johns Hopkins and within the Translational Breast Cancer Research Consortium.
Groups:
- Metastatic Breast Cancer Patients: Adult women with metastatic breast cancer.
Period: Overall Study
Arm/Group | Metastatic Breast Cancer Patients
Started | 182
Completed | 179
Not Completed | 3
Not completed — Physician Decision | 3

BASELINE CHARACTERISTICS:
Arm/Group | Metastatic Breast Cancer Patients
Number analyzed (Participants) | 182
Age, Continuous [Median (Full Range); unit: years] | 56 [28 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 182
  Male | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 182

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival in Patients With a High vs. Low Cumulative Methylation Index (CMI) Value
Time Frame: from week 4 to up to 87 months
Population: 141/179 participants who completed the study were evaluable for this outcome measure. Of these, 8 participants were excluded from analysis for events experienced before week 4, 2 participants had inadequate samples for analysis and data was not collected from 3 participants.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Metastatic Breast Cancer Patients -- CMI High: All subjects enrolled to the study with samples analyzed for the primary objective of DNA methylation in metastatic breast cancer patients who had a high CMI.
- Metastatic Breast Cancer Patients -- CMI Low: All subjects enrolled to the study with samples analyzed for the primary objective of DNA methylation in metastatic breast cancer patients who had a low CMI.
Arm/Group | Metastatic Breast Cancer Patients -- CMI High | Metastatic Breast Cancer Patients -- CMI Low
Number analyzed (Participants) | 71 | 57
months | 2.1 [1.7 to 3.2] | 5.8 [4.7 to 7.4]
Statistical Analysis 1: Comparison: Metastatic Breast Cancer Patients -- CMI High vs Metastatic Breast Cancer Patients -- CMI Low; Test type: Superiority; p = .0002, Gehan; Distributions compared between using the Gehan test, which gives more weight to early differences; Hazard Ratio (HR) = 1.76, 95% CI 2-sided [1.23 to 2.52]

2. Primary Outcome: Changes in Methylated Gene Markers as Measured by Cumulative Methylation Index
Description: log change in cumulative methylation index (CMI) from baseline to week 4. Individual gene methylation (M) is calculated as a methylation index (MI) where MI = (methylated copies)/(number of methylated genes + gene standard copies) * 100. The MI of each sample was averaged across duplicates. The cumulative methylation index (CMI) is the sum of the MI for all genes. The log change from based line to week 4 could increase or decrease. CMI was evaluated as a continuous marker for change from baseline.
Time Frame: baseline, week 4
Population: Data to assess this outcome measure was only collected from 129/182 participants with metastatic breast cancer.
Measure: Mean (Standard Deviation); unit: log CMI change
Arm/Group | Metastatic Breast Cancer Patients
Number analyzed (Participants) | 129
log CMI change | -1.20 (1.84)
Statistical Analysis 1: Comparison: Metastatic Breast Cancer Patients; Hazard ratio; Test type: Other; p = 0.001, Regression, Cox; Cox Proportional Hazard = 1.19, 95% CI 2-sided [1.07 to 1.32]

3. Primary Outcome: Effects of Common Exposures (i.e., Alcohol, Smoking, Medications, and Dietary Factors) on Patterns of Serum Methylation
Time Frame: 9-12 weeks
Population: Data was not collected to assess this outcome measure
Arm/Group | Metastatic Breast Cancer Patients
Number analyzed (Participants) | 0

4. Primary Outcome: Creation of a Predictive Model of DNA Methylation Profiles
Time Frame: 9-12 weeks
Population: Data was not collected to assess this outcome measure
Arm/Group | Metastatic Breast Cancer Patients
Number analyzed (Participants) | 0

5. Secondary Outcome: Overall Survival in Patients With a High vs. Low CMI Value
Time Frame: from week 4 to up to 3 years
Population: 141/179 participants who completed the study were evaluable for this outcome measure. Of these, 7 participants were excluded from analysis for events experienced before week 4, 2 participants had inadequate samples for analysis and data was not collected from 3 participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Metastatic Breast Cancer Patients -- CMI High | Metastatic Breast Cancer Patients -- CMI Low
Number analyzed (Participants) | 62 | 67
months | 12.3 [8.4 to 16.5] | 21.7 [19.3 to 28.3]
Statistical Analysis 1: Comparison: Metastatic Breast Cancer Patients -- CMI High vs Metastatic Breast Cancer Patients -- CMI Low; Test type: Superiority; p = .001, Gehan; Distributions compared between using the Gehan test, which gives more weight to early differences; Hazard Ratio (HR) = 1.70, 95% CI 2-sided [1.18 to 2.45]

6. Secondary Outcome: Correlation of CTCs With Serum Methylation
Time Frame: 3-4 weeks
Population: Data was not collected for this outcome measure
Groups:
- Metastatic Breast Cancer Patients With Measured CMI and CTC: Subjects who had measured values of both CMI and CTC
Arm/Group | Metastatic Breast Cancer Patients With Measured CMI and CTC
Number analyzed (Participants) | 0

7. Other Pre Specified Outcome: Determination if the Addition of CTCs to Serum Methylation Results in an Improved Predictive Model
Time Frame: 3-4 weeks
Reporting Status: Not Posted

8. Post Hoc Outcome: Overall Survival in Participants With High CTC vs. Low CTC
Description: overall survival in participants with high or low cumulative tumor cells (CTC). "high CTC" refers to >5 cells/7.5mL and "low CTC" refers to <5 cells/7.5mL.
Time Frame: 4 weeks
Population: Data for this outcome measure was collected from only 96 participants.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Metastatic Breast Cancer Patients With Measured CTC Values: Subjects with metastatic breast cancer who had measured values of CTC
Arm/Group | Metastatic Breast Cancer Patients With Measured CTC Values
Number analyzed (Participants) | 96
months
  High CTC (>5 cells/7.5 mL) | 8.1 [4.9 to 18.8]
  Low CTC (<5 cells/7.5 mL) | 20.8 [17.5 to 26.6]

ADVERSE EVENTS:
Time Frame: up to 12 weeks from time of consenting to study
Arm/Group | Metastatic Breast Cancer Patients
All-Cause Mortality (participants affected / at risk) | 3/182
Serious Adverse Events (participants affected / at risk) | 3/182
Other Adverse Events (participants affected / at risk) | 0/182
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metastatic Breast Cancer Patients (N=182)
Death (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) — Disease progression NOS

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No